CLINICAL TRIAL: NCT01963845
Title: Sitagliptin Versus Placebo in the Treatment of Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Associate Professor of Clinical Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sitagliptin-NAFLD
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Active drug (Experimental): Sitagliptin 100 mg
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin
  Arms: Active drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) represents a spectrum of diseases ranging from simple steatosis to nonalcoholic steatohepatitis (NASH), the progressive form of liver disease that can lead to cirrhosis and liver-related mortality in persons who drink little or no alcohol. NAFLD is defined as the presence of hepatic steatosis with no evidence of hepatocellular injury in the form of ballooning of the hepatocytes. NASH is defined as the presence of hepatic steatosis and inflammation with hepatocyte injury (ballooning) with or without fibrosis. NASH is benign in many affected individuals but can cause progressive liver injury and, indeed, may be the major cause of cryptogenic cirrhosis1. Currently, there is no FDA approved treatment for NAFLD. Weight loss and exercise are the recommended but often difficult maintain these lifestyle changes in the long term and therefore therapeutic agents have been investigated. In this study, we propose to treat 50 patients with NAFLD and diabetes with either sitagliptin or placebo for 24 weeks. After an initial evaluation for insulin sensitivity and MRI liver fat distribution, patients will receive either 100 mg/day of sitagliptin or placebo. Patients will be monitored at regular intervals for symptoms of liver disease, side effects of sitagliptin and serum biochemical and metabolic indices. At the end of 24-weeks, patients will have a repeat medical evaluation, liver MRI and an optional liver biopsy. Pre and post treatment MRI-derived liver fat content and insulin sensitivity will be compared. The primary end point of successful therapy will be improvement in hepatic steatosis measured by MRI. Secondary end points will be improvement in insulin sensitivity and liver biochemistry.

DETAILED DESCRIPTION:
Primary objectives:

1. To examine the efficacy of sitagliptin 100 mg orally daily versus placebo in improving hepatic steatosis assessed by magnetic resonance imaging in patients with NAFLD.

Secondary objectives:

1. To examine the efficacy of sitagliptin in improving serum AST in patients with NAFLD.
2. To examine the efficacy of sitagliptin in improving serum ALT in patients with NAFLD.
3. To examine the efficacy of sitagliptin in improving serum LDL in patients with NAFLD.
4. To examine the efficacy of sitagliptin in the improvement of insulin sensitivity in patients with NAFLD.

ELIGIBILITY:
44 patients with NAFLD will be randomized to either sitagliptin or placebo for 24-weeks. Enrollment of 50 patients is needed to allow for exclusion of some patients after initial evaluation and a dropout of a small number of patients because of intolerance to sitagliptin.

Inclusion criteria:

1. Age at entry at least 18 years.
2. Serum alanine (ALT) or aspartate (AST) aminotransferase activities that are above the upper limits of normal. 19 or more in women and 30 or more in men.
3. Evidence of hepatic steatosis or liver fat (≥5%) by MRI.
4. Prediabetic patients and controlled diabetic patients as defined by the ADA position statement on diabetes mellitus. Prediabetics have a HbA1c of 5.7 to 6.4 and controlled diabetic patients have an HbA1c between 6.4 and 8.0.
5. Written informed consent.

Exclusion criteria:

1. Uncontrolled diabetes defined as a Hb A1c ≥ 8.0.
2. Evidence of another form of liver disease.

   * Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
   * Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA in serum.
   * Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
   * Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
   * Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
   * Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
   * Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
   * Drug-induced liver disease as defined on the basis of typical exposure and history.
   * Bile duct obstruction as shown by imaging studies.
3. History of excess alcohol ingestion, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1 drink per day: 7 drinks per week) in the previous one year.
4. Advanced liver disease: platelet counts < 75,000/mm3 or prothrombin time >16 seconds or history of bleeding disorders
5. Decompensated liver disease, Child-Pugh score greater than or equal to 7 points
6. History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
7. Recent initiation or change of anti-diabetic drugs, including insulin, sulfonylureas, or thiazolidinediones in the previous 90 days.
8. Use of sitagliptin or other agents in the same class within the 90 days prior to randomization.
9. Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator would preclude treatment with Sitagliptin and adequate follow up.
10. History of acute pancreatitis within the last 5 years with the exception of gallstone pancreatitis.
11. Positive test for anti-HIV.
12. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.
13. Pregnancy or inability to practice adequate contraception in women of childbearing potential.
14. Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study that is suggestive of liver cancer.
15. Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibility hinder completion of the study.
16. Serum creatinine >1.5 mg/dl.
17. Contraindications to Sitagliptin use :

    * History of allergic reaction to Sitagliptin
    * Patients with acute liver injury or unexplained persistent elevations in ALT > 500 U/L at baseline.
    * Women who are pregnant or may become pregnant
    * Nursing mothers
18. Contraindications to MRI:

    * The subject has any contraindication to MR imaging, such as patients with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field.
    * The subject has a history of extreme claustrophobia
    * The subject cannot fit inside the MR scanner cavity

11. RECRUITMENT Enrollment of patients may be initiated once IRB approval is acquired and will continue until June 2015.

Patients will be recruited from the following populations:

* Primary care and internal medicine clinics
* Tertiary referral clinics at the Hillcrest Campus and Perlman Clinics:

  * GI/Liver clinic
  * Liver transplant clinic
  * Obesity clinic
  * Bariatric surgery clinic
  * Diabetes clinic
  * Lipid disorders clinic
* Physicians taking care of the patients would provide information regarding the study and then either refer the patient to our clinic or ask the patient to directly contact the PI or research assistant.
* Patient would be given information regarding possible studies in NAFLD in liver clinic by their providers. We would ask the patient to call or email the PI or research assistant to further discuss the study, if they are interested.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Jan. 1, 2014 to May 1, 2015
Groups:
- Placebo: Sitagliptin-matched placebo tablet
Period: Overall Study
Arm/Group | Placebo | Active Drug
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants] — Subjects recruited from the UCSD hepatology clinic
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 22 | 21 | 43
    >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Liver Fat Relative to Baseline Assessed by MRI-PDFF
Description: Participants liver fat was measured at baseline and 24 weeks. This is the percentage change in liver fat assessed by MRI-PDFF and stratified by treatment group.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percentage change in liver fat
Groups:
- Active Drug: Sitagliptin 100 mg
  Sitagliptin
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 17 | 24
percentage change in liver fat | 13.9 (8.5) | 8.4 (11.6)
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority or Other; p = 0.585, t-test, 2 sided

2. Secondary Outcome: AST, Aspartate Aminotransferase
Description: AST, measured in IU/L at baseline and 24 weeks
Time Frame: Baseline and 24 weeks
Population: All participants with AST measurements at baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 22 | 25
IU/L
  Baseline | 28.5 [19.0 to 37.0] | 28.0 [24.0 to 39.0]
  24 weeks | 23.5 [19.0 to 30.0] | 27.0 [22.0 to 42.0]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Comparison of change in AST values from baseline to 24 weeks between the two groups; Test type: Superiority or Other; p = 0.7583, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: ALT, Alanine Aminotransferase
Description: ALT, measured in IU/L at baseline and 24 weeks
Time Frame: Baseline and 24 weeks
Population: All participants with ALT measurements at baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 22 | 25
IU/L
  Baseline | 40.0 [22.0 to 51.0] | 43.0 [28.0 to 54.0]
  24 weeks | 28.5 [20.0 to 50.0] | 34.0 [27.0 to 56.0]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Comparison of change in ALT values from baseline to 24 weeks between the two groups; Test type: Superiority or Other; p = 0.8569, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: LDL, Low-density Lipoprotein
Description: LDL, measured in mg/dL at baseline and 24 weeks
Time Frame: Baseline and 24 weeks
Population: All participants with LDL measurements at baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 22 | 25
mg/dL
  Baseline | 99.0 [72 to 134] | 100.0 [83.0 to 125.0]
  24 weeks | 101.0 [76.0 to 131.0] | 98.0 [82.0 to 124.5]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Comparison of change in LDL values from baseline to 24 weeks between the two groups; Test type: Superiority or Other; p = 0.7984, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: HOMA-IR, Homeostatic Model Assessment of Insulin Resistance
Description: HOMA-IR, calculated as [(glucose (mg/dL) X insulin (mg/dL)) / 405 ] at baseline and 24 weeks
Time Frame: Baseline and 24 weeks
Population: All participants with HOMA-IR calculated at baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 22 | 25
HOMA-IR score
  Baseline | 5.4 [4.3 to 6.8] | 5.9 [4.4 to 9.2]
  24 weeks | 4.9 [2.9 to 8.9] | 6.8 [4.4 to 9.7]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Comparison of change in HOMA-IR values from baseline to 24 weeks between the two groups; Test type: Superiority or Other; p = 0.5560, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Arm/Group | Placebo | Active Drug
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No